CLINICAL TRIAL: NCT01027507
Title: Relationship Between Postprandial Alterations in Hemodynamics, Blood Pressure, Blood Glucose, Insulin Concentrations, Gastric Emptying, and Satiety
Brief Title: Postprandial Hemodynamics
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Responsible Party: Lars Stavenow, Departments of Medicine, Malmö University Hospital
Other Study IDs: 353/2008b
Record Dates: First submitted 2009-12-07; First posted 2009-12-08 (Estimated); Last update posted 2009-12-08 (Estimated); Status verified 2009-12

CONDITIONS: Heart Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To study the postprandial alterations in hemodynamics and blood pressure in relation to gastric emptying rate, postprandial blood glucose, plasma concentrations of insulin, satiety in healthy subjects.

DETAILED DESCRIPTION:
Ingestion of a meal increase blood flow to the gastrointestinal organs and affects the heart rate, blood pressure, and cardiac output. It is not known through wich mechanisms the heart function changes affects after a meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* history of gastrointestinal disease, abdominal surgery or diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects without symptoms or a history of gastrointestinal disease, abdominal surgery or diabetes mellitus, were included in this crossover study.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2009-01; Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Hlebowicz, MD, PhD, Principal Investigator — Skane University Hospital
Locations (1):
- Departments of Medicine, Malmö University Hospital, Malmo, Sweden

REFERENCES:
- [Derived] Dencker M, Bjorgell O, Hlebowicz J. Effect of food intake on 92 oncological biomarkers by the Proseek Oncology II panel. BMC Res Notes. 2019 Apr 2;12(1):199. doi: 10.1186/s13104-019-4237-9. PMID 30940215
- [Derived] Hlebowicz J, Lindstedt S, Bjorgell O, Dencker M. The effect of endogenously released glucose, insulin, glucagon-like peptide 1, ghrelin on cardiac output, heart rate, stroke volume, and blood pressure. Cardiovasc Ultrasound. 2011 Dec 29;9:43. doi: 10.1186/1476-7120-9-43. PMID 22206473
- [Derived] Hlebowicz J, Lindstedt S, Bjorgell O, Dencker M. Relationship between postprandial changes in cardiac left ventricular function, glucose and insulin concentrations, gastric emptying, and satiety in healthy subjects. Nutr J. 2011 Mar 23;10:26. doi: 10.1186/1475-2891-10-26. PMID 21429209